CLINICAL TRIAL: NCT01022619
Title: The Association Between High Risk Pregnancy and Sleep-disordered Breathing
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Meir Medical Center (Other)
Responsible Party: Isaac Shpirer, MD, head of the sleep laboratory, Asaf Harofeh Medical Center
Other Study IDs: 61/09
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Preeclampsia; Gestational Diabetes; Premature Labor
Keywords: Sleep apnea; high risk pregnancy; fetal outcome; cord blood
MeSH Terms: conditions — Pre-Eclampsia; Diabetes, Gestational; Obstetric Labor, Premature; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cord blood will be obtained in EDTA tubes and serum-seperating tubes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Premature labor: Women at the third trimester of pregnancy with premature contractions and cervical dilation of effacement
- Control: Women at the third trimester of pregnancy with uncomplicated pregnancy
- Pre-eclampsia: Women at the third trimester with pre-eclampsia
- Gestational diabets: Women at the third trimester of pregnancy with gestational diabetes requiring insulin

SUMMARY:
The aim of the present study is to establish, using polysomnographic criteria and prospective nature, whether sleep apnea in pregnancy is more prevalent in women with high risk pregnancies including preeclampsia, gestational diabetes, and pre-mature contractions, and to determine the effect of sleep disordered breathing in pregnancy on fetal outcome. The investigators' hypothesis is that sleep-disordered breathing is more prevalent in women with high risk pregnancy compared to those with uncomplicated pregnancy.

DETAILED DESCRIPTION:
Over the last decade, the association between sleep disordered breathing and pregnancy outcome has been described primarily in case reports. Although recently, larger studies describing adverse pregnancy outcomes in women with sleep disordered breathing has begun to emerge, these studies often lack polysomnographic data and the true prevalence of sleep disordered breathing in pregnancy is not known. We intend to recruit 100 women at the third trimester of pregnancy, who are admitted to the high risk pregnancy unit with pre-eclampsia, gestational diabetes, or premature labor. An additional group of 50 women at the third trimester of an uncomplicated pregnancy will be recruited. All women will fill questionnaires regarding the pregnancy and their sleep and will undergo an overnight sleep study. Women will then be followed until birth. Pregnancy complication, birth and perinatal course will be recorded. Cord blood will be collected from all infants and evaluated for inflammatory cytokines, reactive oxygen species and growth factors. Infants will then be followed for 1 year. Their growth, development and intercurrent illnesses will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 - 39 years
* Over 26 weeks of gestation
* One of the following:

  1. Pre-eclampsia defined as systolic blood pressure > 140 or diastolic blood pressure > 90 and associated proteinuria > 300 mg / 24 h urine collection.
  2. Gestational diabetes requiring insulin treatment
  3. Premature contractions with associated cervical dilation or effacement
  4. Uncomplicated pregnancy

Exclusion Criteria:

* Chronic maternal disease
* Alcohol consumption during pregnancy
* Illicit drug abuse at any time in life
* Fetal abnormalities on obstetric ultrasound

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women in third trimester admitted to the high-risk pregnancy unit and women with uncomplicated pregnancy attending a pre-labor course
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
apnea-hypopnea index | At time of assessment

SECONDARY OUTCOMES:
birth weight, apgar score | at birth
inflammatory markers in cord blood | at birth
growth and development during the 1st year of life | at age 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Shpirer, MD, Principal Investigator — Pulmonary division ans sleep laboratory, Asaf Harofeh Medical Center
Locations (2):
- Israel (2):
  - Meir Hospital, Kfar Saba
  - Asaf Harofeh Medical Center, Ẕerifin